CLINICAL TRIAL: NCT04818827
Title: Ketamine Infusion as Sedative Analgesic in Severe ARDS on Mechanically Ventilated Patients
Brief Title: Ketamine Infusion as Sedative Analgesic in Severe ARDS
Acronym: KISS
Status: Completed | Type: Observational
Sponsor: Interfaith Medical Center (Other)
Responsible Party: Principal Investigator, Ramakanth Pata, Pulmonary Fellow, Interfaith Medical Center
Other Study IDs: KISS 1.0
Record Dates: First submitted 2021-03-19; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Intensive Care Unit Syndrome; Mechanical Ventilation Complication; Sedatives and Hypnotics Causing Adverse Effects in Therapeutic Use; Delirium
Keywords: ketamine; Mechanical ventilation; sedative analgesic; hospital length of stay; Number of ventilator days; mortality
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ketamine group: This cohort includes patients who received ketamine as a sedative analgesic agent during mechanical ventilation
- Non Ketamine group: This cohort includes patients who received sedatives other than ketamine during mechanical ventilation

SUMMARY:
To evaluate whether ketamine is a safe sedative-analgesic agent to be used in an intensive care unit (ICU) setting as compared to traditionally used agents such as propofol, opioids, and midazolam

DETAILED DESCRIPTION:
According to the 2018 Clinical Practice Guidelines for the prevention and management of pain, agitation/sedation, delirium, immobility, and sleep disruption in adult patients in the intensive care unit (ICU), nonbenzodiazepine sedatives (such as propofol and dexmedetomidine) are preferable to benzodiazepine sedatives (such as midazolam and lorazepam) in critically ill, mechanically ventilated patients. Moreover, continuous use of benzodiazepine (more than 48 hours) has been associated with a risk of prolonged sedation and delirium. On the other hand, though propofol has a remarkable safety profile, it carries unfavorable side effects such as dose-dependent hypotension, hypertriglyceridemia, pancreatitis, and propofol syndrome (which is a rare but potentially fatal complication, associated with high-dose propofol infusions, and characterized by severe metabolic acidosis and circulatory collapse).

During the coronavirus disease 2019 (COVID-19) pandemic, an enormous number of patients required mechanical ventilation, which led to the shortage of traditional sedatives such as propofol, dexmedetomidine, midazolam, and lorazepam in the hospitals. In this challenging time, ketamine was used as an alternative sedative infusion. This study is to evaluate whether ketamine is safer compared to other sedatives in severe COVID related ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe acute respiratory distress syndrome (ARDS) due to COVID-19 with an arterial partial pressure of oxygen divided by the inspired oxygen concentration (P/F) ratio < 150 with a minimum 5 cm of positive end-expiratory pressure on a mechanical ventilator

Exclusion Criteria:

* post-cardiac arrest status,
* premorbid diagnosis of dementia,
* dependency on extra-corporeal therapies prior to or during ICU stay

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes patients who are on mechanical ventilators and classified as moderate to severe ARDS with a PF ratio < 150.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-02-14 (Actual)

PRIMARY OUTCOMES:
All-Cause mortality | 10 months (throughout the study period)
  The two groups were compared for all-cause mortality during the ICU stay

SECONDARY OUTCOMES:
Hospital length of stay | 10 months (throughout the study period)
  The two groups were compared for hospital length of stay
Duration of ventilator days | 10 months (throughout the study period)
  The patients in two groups were compared for the duration of ventilator days
Infectious complications | 10 months (throughout the study period)
  The patients in both groups were cultured as clinically suspected for infection. This included blood culture, urine culture and BAL/TTA
Acute Kidney Injury | 10 months (throughout the study period)
  Routine blood samples were obtained that included serum creatinine. Acute kidney injury is defined as per KDIGO
Hemodynamic instability | 10 months (throughout the study period)
  The patients were classified as hemodynamic instability if received vasopressors or ionotropes
Delirium after extubation | 10 months (throughout the study period)
  All patients in the study were routinely screened for delirium using the CAM-ICU score

CONTACTS AND LOCATIONS:
Overall Officials: RAMAKANTH PATA, MD, Principal Investigator — Interfaith Medical Center
Locations (1):
- Interfaith Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Willing to share all aspects of de-identified data
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Available from March 30/2021
Access Criteria: Can be accessed via publishing journal